CLINICAL TRIAL: NCT06295497
Title: Lung Cancer Screening in High Risk NonsmokErs by Artificial InteLligence Device
Brief Title: Lung Cancer Screening by Artificial Intelligence Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Molly SC Li, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LC-SHIELD
Record Dates: First submitted 2024-02-18; First posted 2024-03-06 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Artificial intelligence-based programme (Lung-SIGHT) (Other): Artificial intelligence (AI) algorithms have been demonstrated to function well and complement radiologists as second or concurrent readers in pulmonary nodule detection. AI Lung nodule detection and quantification solution are now widely used in the hospitals in the United Kingdom and at least eight other European countries. The sensitivity of nodule detection by radiologists increased from 72% to 80% with the aid of the AI programme. A clinical trial in Taiwan showed that using AI programme alone achieved an overall sensitivity of 95.6% in nodule detection, and superior performance in detecting nodule sized 4-5 mm comparing to radiologists. Overall, application of AI in CT analysis and lung nodule detection may significantly reduce the cost and workload of radiologist.
  Interventions: Device: Lung-SIGHT

INTERVENTIONS:
Device: Lung-SIGHT — * The LDCT images will be interpreted by an artificial intelligence-based programme (Lung-SIGHT) for lung nodules.
  * LDCT with lung nodules ≥5mm detected by AI programme (AI+) will be sent for reporting by board-certified radiologists.
  * Participants with abnormal LDCT reported by radiologists (Rad+) will be followed up at designated clinic. Management of lung nodules will follow the guidelines below for two years.
  * Participants with negative LDCT determined by AI programme (AI-) will undergo LDCT thorax and blood taking two years later (T1). Patients with lung nodules detected by AI programme (AI+) will be sent for radiologist reporting and those with abnormal CT reported by radiologists (Rad+) will be followed up in lung nodule clinic as per standard of care. Patients with normal second-round LDCT as determined by AI (AI-) or radiologists (AI+ Rad-) do not require follow up.

SUMMARY:
Lung cancer screening is currently not recommended in non-smokers due to paucity of evidence. Emerging evidence suggests that first-degree family history is a strong risk factor for lung cancer in Asian non-smokers. In Asia, lack of resource is a major challenge in successful implementation of lung cancer screening. Artificial intelligence (AI) is a promising tool to overcome this resource. In this study, we aim to study the clinical utility and demonstrate the feasibility of using an AI assisted programme for lung cancer screening in Asian non-smokers with a positive family history. This is a single-arm non-randomized lung cancer screening study. 1000 non-smokers, age 50 to 75 year old, with a first-degree family history of lung cancer, will be enrolled. Participants will undergo low does computed tomography (LDCT) of thorax and blood taking at enrolment. LDCT films will be interpreted by AI softwares for presence of lung nodules. Participants with lung nodules will be further investigated and followed up according to the risk of malignancy. The primary endpoint is the prevalence of early-staged lung cancer detected by first-round LDCT thorax in this population.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all of the following criteria apply:

1. Age 50-75 years old
2. Non-smoker (defined as less than 100 cigarettes in lifetime)
3. Having a first-degree family history of lung cancer
4. Physically fit for curative treatment if early-staged lung cancer is found
5. Able to provide written informed consent
6. Consent to follow up visits and follow up CT scan if indicated
7. Consent to blood taking for translational research

Exclusion Criteria:

Patients who meet any of the following exclusion criteria at screening are not eligible to be enrolled in this study:

1. History of malignancy
2. Smoking history (defined as more than 100 cigarettes in lifetime)
3. Clinical symptoms suspicious for lung cancer e.g. haemoptysis, chest pain, weight loss
4. Medical comorbidities that preclude curative treatment (surgery) for lung cancer, such as severe heart disease, acute or chronic respiratory failure, home oxygen therapy, bleeding disorder
5. Pregnant ladies or ladies planning for conception
6. History of tuberculosis or interstitial lung disease
7. Pneumonia requiring antibiotic treatment within the last 12 weeks
8. CT thorax or chest performed within 2 years (including LDCT or CT coronary angiogram)
9. Unable or unwilling to provide written informed consent

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of early-staged lung cancer detected by first-round LDCT thorax (T0) in a high-risk non-smoker population | 2 years

SECONDARY OUTCOMES:
Sensitivity of AI-assisted programme in lung nodule detection and monitoring compared to radiologist assessment | 2 years
Rate of invasive workup and incidence of associated complications. | 2 years
Prevalence of lung cancer detected by second-round LDCT (T1) in patients with negative first-round LDCT | 2 years
Diagnostic accuracy and discrimination ability of plasma-based fragmentomic assay in detection of lung cancer via assessment of sensitivity, specificity, positive predictive value and negative predictive value | 2 years
To determine the quality adjusted life years (QALYs) gained through screening | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No